CLINICAL TRIAL: NCT07339917
Title: Investigating Predictors of Outcomes From LENS, a Cognitive Bias Modification for Interpretation (CBM-I) Training, in Adults With Elevated Anxiety
Brief Title: Investigating Predictors of Outcomes From LENS
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 363721
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Learning Effective New Strategies (LENS) — Learning Effective New Strategies (LENS) is a Class I digital mental health intervention developed by King's College London, of which the overall purpose is to shift the way people think about ambiguous situations to be more positive and helpful. LENS achieves this through a drill-like training where users are prompted to visualise positive conclusions to numerous situations which are ambiguous and could be interpreted in either negative or positive ways. This training involves completing 12 sessions over 4 weeks. This type of training is known as cognitive bias modification for interpretation bias (CBM-I), which trains individuals to think in a more positive, adaptive way. The intended use of LENS is to reduce anxiety, depression and/or repetitive negative thinking in individuals with anxiety (low to high levels), depression (low to moderate levels), and/or repetitive negative thinking (moderate to high levels).

SUMMARY:
Anxiety is a very common mental health problem. For people living with anxiety, it can have a huge impact on their lives. There are treatments that can help, such as Cognitive Behavioural Therapy (CBT). However, about half of the people who receive treatment still struggle with anxiety after treatment is complete, and we do not yet know why. In this study, we hope to find factors that help explain why people respond differently to anxiety treatment. To answer this question, people in this study will receive a digital anxiety treatment called Learning Effective New Strategies (LENS). LENS is a type of brain training that helps people make less negative interpretations of uncertain situations and information. LENS has been proven to help reduce worry and anxiety, and improve mood (Hirsch et al., 2021). After participants finish LENS, we will measure how their patterns of thinking and mood changes over treatment and during the following five months. We will invite people to take part through multiple existing research studies (e.g. GLAD, TEDS) who have already shared their genetic data (information about their DNA). This way of recruiting would allow us to combine this genetic data with information from questionnaires to look for genetic and psychological factors that are linked with how well someone's anxiety improves after treatment. This research could help us understand what factors are linked to a person's outcomes from treatment. In the future, this could help health professionals personalise anxiety treatment and offer the right treatment to people sooner. This would mean that fewer people need to try multiple treatments before finding one that works. We hope this study will improve care for people living with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18
* Fluent in English
* Normal or corrected to normal hearing
* Normal or corrected to normal vision
* Currently experiencing anxiety (GAD-7 score ≥ 8)
* Access to stable internet connection
* Access to smartphone, laptop, computer, or tablet

Exclusion Criteria:

* Current high levels of suicidal ideation, as defined by a score ≥ 2 on Item 9 of the PHQ-9 OR score of 1 on Item 9 of the PHQ-9 and score ≥21 on the SIDAS
* Suicide attempt in past two years.
* Current or history of psychosis or bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have taken part in previous genetic cohort studies, namely GLAD, TEDS and Genes & Health, will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4400 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2032-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder-7 score | 8 week follow up
  General Anxiety Disorder-7 score on GAD-7 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Colette R Hirsch, Principal Investigator — King's College London; Thalia Eley, Principal Investigator — King's College London; Gerome Breen, Principal Investigator — King's College London; Ewan Carr, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided